CLINICAL TRIAL: NCT00986518
Title: Controlled and Selective Depletion of Regulatory T-cell for Cancer Treatment, Efficacy and Safety Study
Brief Title: T Regulatory Lymphocytes (Treg) Depletion for Cancer Treatment Efficacy and Safety Study
Acronym: STARTREK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P080601
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: Advanced Colorectal Cancer; Hepatic and/or lung metastasis; Adaptive autologous cell immunotherapy; T- regulatory lymphocyte depletion; Neo-adjuvant reduced intensity chemotherapeutic conditioning
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adaptive cell immunotherapy (Experimental)
  Interventions: Biological: Adaptive autologous cell immunotherapy

INTERVENTIONS:
Biological: Adaptive autologous cell immunotherapy — each patient will undergo a blood cytapheresis to collect circulating lymphocytes. Ex-vivo cell sorting procedure will deplete patient's collected lymphocytes from regulatory T cells. Autologous Treg-depleted lymphocytes will be administered to the patient following a 5-day reduced intensity chemo-therapeutic conditioning.

SUMMARY:
T regulatory lymphocytes were shown to be partly responsible for immune tolerance to cancer cells. In that respect these cells oppose to the mounting of an efficacious immune response needed to cure cancer. To treat advanced metastatic colorectal cancer, the investigators propose an immunotherapy consisting in autologous lymphocytes infusion depleted from T-regulatory cells, associated with a 5-day prior lymphoid-ablative chemotherapy associating cyclophosphamide (day 1 & 2) with fludarabine (day 1 to 5). To administer treatment and monitor chemotherapy safety, patients will be hospitalized for 3 weeks until complete recovery from chemotherapy. Patients will then be followed-up ambulatory for 9 months during which time they will be assessed for tumor size with computed tomography (CT) - scan (primary criteria).

DETAILED DESCRIPTION:
The primary goal of the proposed clinical trial is to eliminate cancer tumor using an autologous cell therapy aiming at mounting an efficient immune anti-tumor response by selectively depleting regulatory T-cell during a controlled amount of time. This strategy will be tested in patients with hepatic metastases from colorectal who are not eligible for surgery.

This is an open-label single cohort phase I-II therapeutic trial. Patients with hepatic metastases from primary colorectal cancer, not eligible to surgery and relapsing from conventional chemotherapy and/or targeted therapy, will be included.

Following patient inclusion:

1. A lymphapheresis will be performed at D-15 which will be subjected to cell sorting /purification of regulatory T cells on the one hand and T lymphocytes depleted from regulatory T cells (effectors T-cells) on the other, and subsequently frozen and stored (The procedures for ex vivo regulatory T cell depletion has been validated in a previous study - AFSSAPS- TC 192) ;
2. A lymphoid-ablative chemotherapy (cyclophosphamide + fludarabine) will be perform from D1 to D5,
3. Autologous effector T-cells administration will be performed at D7. Efficacy will be assessed through tumor size change. Change in tumor size will be assessed with CTscans (RECIST criteria), MRIs (functional criteria following injection: DCEMRI and diffusion MRI to assess change in cellularity and tumor necrosis and morphological criteria RECIST), and sonography with contrast injection (to assess vascular microcirculation). Assessments will be done prior to lymphoid-ablation and then monthly for 9 months. Safety will be systematically assessed daily during in-patient period using the World Health Organisation - Common Toxicity Criteria (WHO-CTC).

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal adenocarcinoma histologically proven;
* Hepatic or lung metastasis (at least one with size >1cm on CT-scan);
* Not eligible for surgery;
* Prior treatment with fluoropyrimidines, CPT11, oxaliplatine and EGFR antibodies (Cetuximab ou Panitumumab) ± bevacizumab; When tumor has a mutated Kras, prior treatment with EGFR antibodies is not mandatory;
* No local recurrence (on CT-scan, sonogram and/or colonoscopy);
* Karnofsky index > 70 and PS 0 or 1;
* ASA Score < 3 ;
* Absence of chronic hepatopathy ;
* Lab test : WBC: neutrophil> 2.0 109 / l, lymphocytes > 1.5 109 / l; creatinine < 1.5 x ULN or clearance ≥ 60 ml/min; AST et ALT< 5 x ULN, alkaline phosphatases < 3 x ULN; LDH < 3 x ULN; negative Coombs test ;
* Signed informed consent.

Exclusion Criteria:

* Peritoneal carcinosis on CT-scan, MRI or PET-scan;
* Contra-indication to MRI;
* Patient with known allergy to iodinated contrast agent, gadolinium or Sulfate Hexafluoron ;
* Presence of metastasis at sites other than lung and liver;
* Documented history of auto-immune disease and/ or progressing disease;
* Infection at whatever site;
* Documented history of allo- or autograft;
* Undernutrition, BMI < 18;
* History of other cancer < 5 years (excluding cancer in situ of the cervix and baso-cellular tumor of the skin) or progressing disease;
* Women of child bearing age without contraception , or pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Tumor size of hepatic and/or lung metastases, as measured with tomodensitometry (RECIST 1.1 criteria) | from Month 1 to Month 9

SECONDARY OUTCOMES:
MRI : Assessment of tumor necrosis, cellularity and morphological criteria RECIST 1.1 (functional criteria following injection : DCEMRI and diffusion MRI) | Month 1 to Month 9
Sonography : assessment of vascular micro-circulation with contrast injection, | Month 1 to Month 9
Immune cell reconstitution will be assessed through measuring rate of regulatory T-cell reconstitution, | day 7 to 28
Clinical Exam (WHO-CTC), Vital Signs, Adverse events | day 1 to 28
Laboratory test: hepatic function, immune function, haematology | day 1 to 28

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Service hépato-gastro-enterologie, Pitié-Salpêtrière Hospital, Paris, France